CLINICAL TRIAL: NCT06786403
Title: Investigating the Effectiveness of the Supplement Containing Enteric-coated Bromelain (Anaheal 1200 GDU) in Healing Wounds, Pain, and Inflammation in Patients Over 18 Years Old with Diabetic Foot Ulcers Compared to Placebo
Brief Title: The Effects of Bromelain Supplement in Patients with Diabetic Foot Ulcers
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Dr Azita Hekmatdoost (Other)
Responsible Party: Sponsor-Investigator, Dr Azita Hekmatdoost, Professor, National Nutrition and Food Technology Institute
Organization: National Nutrition and Food Technology Institute (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 162948239
Record Dates: First submitted 2025-01-15; First posted 2025-01-22 (Actual); Last update posted 2025-01-22 (Actual); Status verified 2025-01

CONDITIONS: Diabetic Foot Ulcer (DFU)
Keywords: diabetic foot ulcer; bromelain
MeSH Terms: conditions — Diabetic Foot | interventions — Bromelains

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- placebo (Placebo Comparator): placebo
  Interventions: Dietary Supplement: Placebo
- enteric-coated bromelain (Active Comparator): Intervention : Bromelain
  Interventions: Dietary Supplement: Bromelain

INTERVENTIONS:
Dietary Supplement: Bromelain — Dietary Supplement: Bromelain 1000 mg/day
  Arms: enteric-coated bromelain
Dietary Supplement: Placebo — Placebo (1000 mg/day)
  Arms: placebo

SUMMARY:
This study will be conducted on people over 18 with diabetic foot ulcers.. The first group will receive the standard treatment along with bromelain supplement and the second group will receive the standard treatment and placebo. The informed consent form prepared in advance will also be provided to the patients so that they are fully familiar with the study process. Wound surface area, rate of pain, rate of inflammatory factors (ESR and CRP) will be assessed at baseline and every two weeks.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years old
* Patients diagnosed with diabetic foot ulcers of category 0, 1 and 2 according to the Wagner criteria
* Patients aware of the study process for monitoring after filling out the informed consent form

Exclusion Criteria:

* People who are allergic to pineapple, celery, carrot and fennel
* Pregnant and lactating women
* Severe kidney failure (GFR<30)
* Severe liver failure (Child Pugh B, C)
* Patients with hemophilia
* People taking anticoagulant drugs, anti-platelet and thrombolytic
* Patients with irregular heartbeat and tachycardia
* Patients with asthma

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2025-03 (Estimated); Primary Completion 2025-08 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
Wound surface area | At baseline and every 2 weeks until the end of treatment at 8 weeks
  Dimensions (length and width) by Image J

SECONDARY OUTCOMES:
The amount of pain | At baseline and every 2 weeks until the end of treatment at 8 weeks
  By Visual Analogue Scale (VAS)
The amount of inflammation | At baseline and every 4 weeks until the end of treatment at 8 weeks
  Lab test parameters of ESR & CRP

CONTACTS AND LOCATIONS:
Overall Officials: Mobina Tajdari, PharmD Student, Principal Investigator; Kamyab Andarzbakhsh, PharmD, Principal Investigator
Locations (1):
- Iran, Tehran, Tehran Province, Iran

IPD SHARING:
Plan to Share IPD: Undecided